CLINICAL TRIAL: NCT07394192
Title: Exploratory Study on the Efficacy and Safety of Short-Course Radiotherapy With Tumor-Draining Lymph Node Preservation Followed by PD-1 Inhibitors in pMMR/MSS Stage II-III Rectal Cancer
Brief Title: Short-Course Radiotherapy With Tumor-Draining Lymph Node Preservation Followed by PD-1 Inhibitors in pMMR/MSS Stage II-III Rectal Cancer
Acronym: PKUCH- R11
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PKUCH- R11
Record Dates: First submitted 2026-01-18; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Rectal Cancer; Radiotherapy; PD-1 Inhibitor
Keywords: short-course radiotherapy; tumor-draining lymph nodes; PD-1 inhibitors; pMMR/MSS; locally advanced rectal cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental arm (Experimental): Neoadjuvant therapy with short-course radiotherapy that preserves tumor-draining lymph nodes, followed by 4 cycles of PD-1 inhibitors
  Interventions: Radiation: short-course radiotherapy that preserves tumor-draining lymph nodes

INTERVENTIONS:
Radiation: short-course radiotherapy that preserves tumor-draining lymph nodes — Patients with stage II-III pMMR/MSS locally advanced rectal cancer receive neoadjuvant therapy with short-course radiotherapy that preserves tumor-draining lymph nodes, followed by 4 cycles of PD-1 inhibitors

SUMMARY:
This study aims to evaluate the efficacy (pathological complete response rate) of short-course radiotherapy with preservation of tumor-draining lymph nodes followed by sequential PD-1 inhibitor neoadjuvant therapy in patients with stage II-III pMMR/MSS locally advanced rectal cancer.

DETAILED DESCRIPTION:
This study is a single-arm, open-label exploratory clinical trial designed to investigate the feasibility and preliminary efficacy of a novel neoadjuvant treatment strategy for locally advanced rectal cancer. The strategy combines short-course radiotherapy (SCRT) with deliberate preservation of tumor-draining lymph nodes, followed by sequential PD-1 inhibitor therapy, with the aim of enhancing antitumor immune activation prior to definitive surgery. Given the exploratory nature of the study, no blinding will be applied, and both investigators and participants will be aware of the assigned treatment. Approximately 44 eligible patients are planned for enrollment.

The study is conducted across four sequential phases: screening and enrollment, neoadjuvant treatment, surgical intervention, and postoperative follow-up. During the screening phase, eligibility will be confirmed through histopathological evaluation, molecular testing, and standardized imaging assessments to establish disease stage and anatomical suitability for the protocol-defined treatment approach.

Neoadjuvant treatment begins with short-course radiotherapy administered in the first week after enrollment. Radiotherapy will be delivered using volumetric modulated arc therapy (VMAT) following standard procedures for patient positioning, immobilization, CT/MRI simulation, target volume delineation, treatment planning, and image-guided verification. In contrast to conventional pelvic irradiation, the clinical target volume is intentionally limited to the primary rectal tumor, excluding tumor-draining lymph nodes and elective pelvic nodal regions, in order to preserve regional immune structures. The prescribed dose is 25 Gy delivered in five fractions over five consecutive working days. Patients will be closely monitored for acute radiation-related toxicities, which will be graded and managed according to standard criteria.

Two weeks after completion of radiotherapy, patients will initiate immunotherapy. Sintilimab, a PD-1 inhibitor, will be administered intravenously at a fixed dose of 200 mg every three weeks for four cycles. Prior to each cycle, patients will undergo routine safety evaluations, including physical examination and laboratory testing, to assess treatment tolerance and determine eligibility for continued dosing. Treatment interruption, delay, or discontinuation will be guided by protocol-defined toxicity management rules.

A comprehensive restaging assessment will be performed approximately 2-4 weeks after completion of neoadjuvant therapy using standardized imaging modalities, including pelvic MRI and thoracoabdominal CT. Patients without evidence of disease progression will proceed to definitive surgical management. Radical resection with total mesorectal excision (TME) is required, with the specific surgical procedure selected according to tumor characteristics and individual clinical considerations.

Postoperative management will be determined based on pathological findings and multidisciplinary team discussion approximately one month after surgery. All patients will then enter a structured follow-up program lasting three years, with visits scheduled every three months. Follow-up evaluations will focus on disease status, survival outcomes, and the assessment of late treatment-related toxicities, using clinical examinations, laboratory tests, tumor markers, and imaging studies as clinically indicated.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old, regardless of sex.

  * Fibrocolonoscopy or digital rectal examination indicates that the distal border of the lesion is located 5-10 cm from the anal verge.

    * Pathologically confirmed rectal adenocarcinoma.

      * Imaging examinations (including pelvic MRI and chest-abdominal CT) confirm a clinical stage of II/III (cT3-T4aN0 or cT2-4aN+, MRF (-), with no distant metastasis) according to the AJCC Cancer Staging Manual, 8th Edition (2018) (for detailed TNM staging of rectal cancer).

        * If N+, metastatic lymph nodes are confined to the mesorectal and superior rectal artery drainage regions, with no lateral pelvic lymph node metastasis.

          ⑥ Confirmed by immunohistochemistry or molecular testing to be mismatch repair proficient (pMMR) or microsatellite stable (MSS).

          ⑦ Eastern Cooperative Oncology Group (ECOG) Performance Status score of 0-1 (see Appendix 2 for details).

          ⑧ Meeting the following laboratory criteria: Hemoglobin ≥ 90 g/L, white blood cell count ≥ 3.5 × 10⁹/L; Neutrophil count ≥ 1.5 × 10⁹/L, platelet count ≥ 100 × 10⁹/L; Creatinine ≤ 1.0 × upper limit of normal (ULN), blood urea nitrogen (BUN) ≤ 1.0 × ULN; Alanine aminotransferase (ALT) ≤ 1.5 × ULN; Aspartate aminotransferase (AST) ≤ 1.5 × ULN; Alkaline phosphatase (ALP) ≤ 1.5 × ULN; Total bilirubin (TBIL) ≤ 1.5 × ULN; Urine protein negative; normal coagulation time; normal thyroid function.

          ⑨ Patients with primary rectal cancer must have undergone no surgical interventions (excluding palliative stoma formation), chemotherapy, or other antitumor treatments from the time of diagnosis to enrollment.

          ⑩ The planned radiation field must have no history of prior radiotherapy.
          * The patient voluntarily agrees to participate in this study, signs the informed consent form, demonstrates good compliance, and is willing to cooperate with follow-up visits and data provision.

Exclusion Criteria:

* Previous treatment with anti-PD-1/L1, anti-CTLA-4 immunotherapies, or other investigational immunotherapeutic agents is excluded.

  * Patients with severe autoimmune diseases are excluded, including active inflammatory bowel disease (such as Crohn's disease, ulcerative colitis), rheumatoid arthritis, scleroderma, systemic lupus erythematosus, autoimmune vasculitis (e.g., Wegener's granulomatosis), etc.

    * Patients with symptomatic interstitial lung disease or active infectious/non-infectious pneumonitis are excluded.

      * Patients with clinical or imaging evidence of intestinal obstruction or perforation, or those deemed by the investigator to be at high risk of perforation or hemorrhage, are excluded.

        * History of other malignancies, excluding curatively treated non-melanoma skin cancer and carcinoma in situ of the cervix, are excluded.

          * Patients with severe cardiovascular or cerebrovascular diseases are excluded, including cerebrovascular accidents, transient ischemic attacks, myocardial infarction within 6 months prior to enrollment, or significant vascular diseases (including but not limited to aortic aneurysms requiring surgical repair or recent arterial thrombosis). Also excluded are those with poorly controlled cardiac symptoms or conditions, such as unstable angina, heart failure of New York Heart Association (NYHA) Class II or higher, left ventricular ejection fraction (LVEF) < 50% on echocardiography, or severe arrhythmias uncontrolled by medication.

            * Physical examination findings, clinical laboratory abnormalities, or other uncontrolled conditions that, in the investigator's judgment, may interfere with the study results or increase the patient's risk of treatment complications are excluded.

              * Lactating or pregnant women are excluded. ⑨ Patients with congenital or acquired immunodeficiency diseases, including human immunodeficiency virus (HIV) infection, or a history of organ transplantation or allogeneic stem cell transplantation, are excluded.

                ⑩ Known active hepatitis B virus (HBV) infection, hepatitis C virus (HCV) infection, or active tuberculosis are excluded.

                ⑪ Patients with concurrent use of other immunomodulators, chemotherapeutic agents, other investigational drugs, or requiring long-term corticosteroid therapy are excluded.

                ⑫ Patients with psychiatric disorders, substance abuse, or social issues that may affect compliance, as determined upon physician review, are excluded.

                ⑬ Patients with allergies or contraindications to the investigational drug(s) are excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2031-12-31 (Estimated)

PRIMARY OUTCOMES:
pathologic complete response rate | Perioperative
  Defined as the absence of residual tumor cells in the surgically resected specimen after neoadjuvant therapy, including both the primary site and lymph nodes.

SECONDARY OUTCOMES:
tumor regression grade | Perioperative
  The extent of postoperative tumor regression is graded and assessed according to the American Joint Committee on Cancer (AJCC) criteria, and the proportions of different grades are calculated.
R0 Resection Rate | Perioperative
  R0 Resection Rate is defined as the proportion of patients in whom a complete microscopic resection is achieved. Specifically, it indicates that no residual tumor cells are found at the microscopic level on the surgical margin after pathological examination of the resected specimen, also known as a negative microscopic margin.
30-Day Postoperative Complication Rate | within the first 30 days after the operation
  30-Day Postoperative Complication Rate is defined as the proportion of patients who experience one or more adverse events directly related to the surgical procedure within the first 30 days after the operation, with the severity of each complication classified according to the Clavien-Dindo Classification system.
3-Year Local-Regional Recurrence Rate | 3 years following surgery
  The cumulative incidence of disease recurrence confined to the primary tumor site (local) and/or the regional lymph node basins, assessed at 3 years following surgery. This rate is typically estimated using the Kaplan-Meier method.
3-Year Distant Metastasis Rate | 3 years following the surgery
  The cumulative incidence of cancer spread to distant organs or sites beyond the primary tumor region and its local lymphatic drainage area, assessed at 3 years following the surgery. This rate is typically estimated using the Kaplan-Meier method.
3-Year Disease-Free Survival (DFS) Rate | 3 years following surgery
  The proportion of patients who remain alive and free from any documented recurrence (local, regional, or distant), secondary primary cancer, or death from any cause, assessed at 3 years following surgery. The rate is estimated using the Kaplan-Meier method.
3-Year Overall Survival (OS) Rate | 3 years following surgery.
  The proportion of patients who are still alive from any cause, assessed at 3 years following surgery. This rate is estimated using the Kaplan-Meier method.
Toxicity Profile During Neoadjuvant Therapy (Graded by CTCAE v5.0) | From the initiation of neoadjuvant therapy until 90 days after the last dose
  The occurrence and severity of adverse events (toxicities) during the neoadjuvant treatment period will be documented and graded according to the Common Terminology Criteria for Adverse Events (CTCAE), Version 5.0.
EORTC QLQ-C30 questionnaire score | Baseline and very 3 months postoperatively until 3 years
  The impact of treatment on patients' quality of life (assessed using the EORTC QLQ-C30 questionnaires)
EORTC QLQ-CR29 questionnaire score | Baseline and very 3 months postoperatively until 3 years
  The impact of treatment on patients' quality of life (assessed using the EORTC QLQ-CR29 questionnaires)
the Low Anterior Resection Syndrome score | Baseline and very 3 months postoperatively until 3 years
  The impact of treatment on patients' anorectal function (evaluated with the Low Anterior Resection Syndrome score questionnaire)

IPD SHARING:
Plan to Share IPD: No